CLINICAL TRIAL: NCT06518538
Title: A Phase 2 Single Center Open-Label Trial to Evaluate Efficacy and Safety of Devimistat in Combination With Modified FOLFIRINOX (mFFX) in 2nd Line Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Evaluate Efficacy of Devimistat in Combination With mFFX in 2nd Line Patients With Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: due to study redesign
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC004
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer Stage IV
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613+mFFX (Experimental): Day 1: Devimistat at 500 mg/m2 IV infusion over 2 hours mFFX (given immediately after devimistat administration):
  * Oxaliplatin at 60 mg/m2 given as a 2-hr IV infusion
  * Folinic acid at 400 mg/m2 given as 30- 90 min infusion immediately after oxaliplatin, and concurrently with Irinotecan at 120 mg/m2 given as a 90-min ( IV infusion via a Y-connector.
  * Fluorouracil (5-FU) 42-48-hr infusion at 2,200 mg/m2, starting immediately after completion of folinic acid and irinotecan
  Day 2:
  mFFX:
  ▪ Completing the remaining of the 5-FU 42-48-hr infusion starting on day 1
  Day3:
  mFFX: ▪ Completing the remaining of the 5-FU 42-48-hr infusion starting on day 1, 2 and disconnect the 5-FU pump
  Devimistat:
  ▪ Devimistat (500 mg/m2), IV infusion over 2 hours via a central venous catheter after completion of 5-FU infusion.
  Day 8:
  Devimistat (500 mg/m2), IV infusion over 2 hours via a central venous catheter
  Interventions: Drug: CPI-613, modified Folfirinox

INTERVENTIONS:
Drug: CPI-613, modified Folfirinox — * CPI-613, devimistat
  * mFFX: Oxaliplatin, Folinic acid, Fluorouracil and Irinotecan

SUMMARY:
Open label, randomized phase II study to evaluate efficacy and safety of CPI-613 + mFFX in patients with metastatic adenocarcinoma of the pancreas with age range of 18 to 75 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic stage IV adenocarcinoma of the pancreas
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Male and female patients 18 - 75 years of age
* Measurable disease determined using guidelines of Response Evaluation Criteria In Solid Tumors (RECIST version 1.1)
* Recurrrence or progression while on FFX therapy.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must agree to use acceptable highly effective contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive(s), intrauterine hormone releasing system (IUS), bilateral tubal occlusion or vasectomized partner) during and for 6 months after last study dose and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Males with female partners (of childbearing potential) and female partners (of childbearing potential) with male partners must agree to use double barrier contraceptive measure (a combination of male condom with either cap, diaphragm or sponge with spermicide) in addition to oral contraception, or avoidance of intercourse during the study and for 6 months after last study dose is received
* At least 4 weeks from major surgery with resolution of any sequela to date of enrollment
* Laboratory values ≤2 weeks during screening must be:
* Adequate hematologic values

  * Platelet count ≥100,000 cells/mm3 or ≥100 bil/L;
  * Absolute neutrophil count [ANC] ≥1,500 cells/mm3 or ≥1.5 bil/L;
  * Hemoglobin >9 g/dL or >90 g/L
* Adequate hepatic function

  * Aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL] (≤5xUNL if liver metastasis present)
  * Alanine aminotransferase [ALT/SGPT] ≤3x UNL (≤5x UNL if liver metastasis present)
  * Bilirubin (≤1.5x UNL); bilirubin ≤ 2.5 x ULN for subjects with Gilbert's syndrome
* Adequate renal function

  * Serum creatinine clearance CLcr > 30 mL/min). (Cockcroft-Gault Formula should be used for CrCl calculation)
* Adequate coagulation function

  * International Normalized Ratio or INR must be <1.5 unless on anticoagulants
* No evidence of active infection and no serious infection within the past 30 days. Patient must have completed antibiotic course.
* Mentally competent, ability to understand and willingness to sign the informed consent form and follow protocol requirements

Exclusion Criteria:

* Endocrine or acinar pancreatic carcinoma
* Known cerebral metastasis, central nervous system (CNS), or epidural tumor
* Patients with hypersensitivity to devimistat, FFX treatment or any of their excipients
* Patients receiving any other investigational systemic agent for any indication within the past 2 weeks prior to initiation of devimistat treatment
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., Hemophilia A)
* Female patients who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after the last dose of study treatment
* Female patients of childbearing potential with a positive pregnancy test assessed by a serum pregnancy test at screening
* Male patients unwilling to abstain from donating sperm during treatment and for 6 months after completion of study treatment
* Active heart disease including but not limited to symptomatic congestive heart failure (NYHA class 3 or 4), symptomatic coronary artery disease, symptomatic angina pectoris, or symptomatic myocardial infarction
* Patients with a history of myocardial infarction that is <3 months prior to registration
* Prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, in situ cancer, localized prostate cancer (Gleason score <8), or adequately treated cancer from which the patient has been disease-free for at least 3 years prior to screening
* Unwilling or unable to avoid the concomitant use of strong CYP3A4 inducers or inhibitors during treatment with irinotecan (Listed in the APPENDIX II: CYP3A4 Inducers or Inhibitors)
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 470 milliseconds (ms) (CTCAE grade 1) using Fridericia's QT correction formula (i.e. QTcF)
* A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
* The use of concomitant medications except anti-emetics that prolong the QT/QTc intervals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) [Time Frame: At least 2 months (minimum of 4 cycles)] Defined as the rate of Complete Response (CR) plus Partial Response (PR) | 12 months

SECONDARY OUTCOMES:
Overall Survival (OS) Defined as the duration from the date of randomization to the date of death from any cause | 24 months
Progression Free Survival (PFS) Defined as the duration from the date of randomization to the date of progressive defined as the duration from the date of randomization to the date of progressive disease or death from any cause. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hirschfeld Oncology, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided